CLINICAL TRIAL: NCT02198638
Title: Influenza Vaccination of HCW and Hospital Acquired Influenza in Patients
Brief Title: Effect of Influenza Vaccination of Healthcare Workers (HCW) on the Risk of Influenza in Patients Hospitalized in Short Stays Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013.814; 2012-A01503-40 (Other: (N°ID-RCB) France: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2014-07-15; First posted 2014-07-23 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Patient With Influenza Like Illness
Keywords: Influenza; Vaccination rate; Hospital acquired infection
MeSH Terms: conditions — Influenza, Human; Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients or healthcare workers (Other)
  Interventions: Biological: A nasal swab

INTERVENTIONS:
Biological: A nasal swab — A nasal swab was performed by a research assistant and influenza virus infection was confirmed by enzyme-linked immunosorbent assay and reverse transcription-polymerase chain reaction on viral cultures

SUMMARY:
Hospital acquired influenza is associated with significant morbidity and mortality in hospitalized patients notably elderly patients. Vaccination of HCW is recommended to prevent influenza transmission in healthcare setting.

Outbreaks of hospital acquired influenza were reported in stays with high vaccine coverage in patients (higher than 85%). It is necessary to underline that an adequate vaccine cover in the elderly population will not necessarily result in a total control of the incidence. Consequently, the prevention of influenza outbreaks in this vulnerable population must also include the reduction of the exposure to the influenza viruses, in particular thanks to the vaccination of HCW.

A pilote case-control study, implemented in Edouard Herriot hospital (at Lyon University hospitals), indicates that a shielding effect of more than 35% of vaccinated HCW on hospital acquired influenza among patients (Bénet et al.; BMC Infectious Diseases 2012). The results suggest a protective effect but investigations, carried out on a more important sample are needed to validate the benefit of HCW vaccination.

The aim of this prospective multicentric cohort study is to estimate incidence of influenza among hospitalized patients according to % of influenza vaccination of HCW in short stay units.

ELIGIBILITY:
Inclusion Criteria:

* All adults patients and healthcare workers of the participating units
* With Influenza Like Illness

Exclusion Criteria:

* Patients aged < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Incidence of influenza among hospitalized patients according to % of influenza vaccination of HCW in short stay units | After 16 months (2 influenza seasons: from 15 December 2013 to 15 April 2014 and from 15 December 2014 to 15 April 2015)
  Study participation was proposed to each patient who presented ILI (influenza like illness) at admission or during hospitalization. ILI was defined as fever >37.8°C or cough or sore throat. Vaccination against influenza during the ILI season was collected by oral interview. After the interview, a nasal swab was performed by a research assistant and influenza virus infection was confirmed by enzyme-linked immunosorbent assay and reverse transcription-polymerase chain reaction on viral cultures.

SECONDARY OUTCOMES:
Estimation of influenza vaccine failure according to serotyping of viral strains | After 16 months (2 influenza seasons: from 15 December 2013 to 15 April 2014 and from 15 December 2014 to 15 April 2015)
  strains of confirmed influenza virus were analysed by reverse transcription-polymerase chain reaction on viral cultures.
Does incidence of community influenza influence hospital acquired influenza infections | After 16 months (2 influenza seasons: from 15 December 2013 to 15 April 2014 and from 15 December 2014 to 15 April 2015)
  comparison of results observed during the 2 seasons

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hospices Civils de Lyon - Hôpital Edouard Herriot, Lyon
  - Centre Hospitalier Universitaire - Saint Etienne, Saint-Etienne

REFERENCES:
- [Result] Amour S, Benet T, Regis C, Robert O, Fontana L, Lina B, Pozzetto B, Berthelot P, Vanhems P. Effect of influenza vaccination among healthcare workers on hospital-acquired influenza in short-stay hospitalized patients: A multicenter pilot study in France. Infect Control Hosp Epidemiol. 2022 Dec;43(12):1828-1832. doi: 10.1017/ice.2022.68. Epub 2022 Apr 6. PMID 35382916